CLINICAL TRIAL: NCT05051800
Title: Enhancing Coping and Communication in Children With Cancer and Their Parents: A Novel Internet Intervention
Brief Title: Enhancing Coping and Communication in Children With Cancer and Their Parents
Acronym: ALSF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment of participants was interrupted by the COVID-19 pandemic and the funding for the study ended before the targeted enrollment could be completed.
Sponsor: Vanderbilt University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Bruce Compas, Patricia and Rodes Hart Professor, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 170111
Record Dates: First submitted 2019-06-18; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Pediatric Cancer
Keywords: Pediatric cancer; Coping
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Recruitment and randomization of participants into an online support program vs. usual care. Participants in the usual care condition offered the program after 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention (Experimental): Families will receive the online program to support coping and communication near the time of a child's cancer diagnosis
  Interventions: Behavioral: Online Program to Support Coping and Communication in Families
- Delayed Intervention (Active Comparator): Families will receive the online program to support coping and communication approximately 6 months after a child's cancer diagnosis
  Interventions: Behavioral: Online Program to Support Coping and Communication in Families

INTERVENTIONS:
Behavioral: Online Program to Support Coping and Communication in Families — Parents and children will access online materials designed to support the use of effective ways to cope with the diagnosis and treatment of cancer and to support open and communication.

SUMMARY:
Childhood cancer patients and their parents are faced with significant stress at the time of diagnosis, during treatment, and over the course of recovery. The stress of cancer and its treatment can lead to significant emotional distress for many families. However, most families do not have access to programs that offer support for coping with cancer-related stress. The proposed work will address this gap by testing of the possible benefits of a novel internet delivered program to support children with cancer and their parents in coping with and communicating about a child's cancer. The research team includes experts from Vanderbilt University and Nationwide Children's Hospital with experience in pediatric oncology; stress, coping, and family communication in pediatric cancer; internet interventions in pediatric populations; and family-focused interventions to build coping and parenting skills. The study will test the effects of this program in 150 families of children with newly diagnosed cancer on reducing emotional distress up to 12 months after participation in the program. This project has the potential to lead to an evidence-based program to improve quality of life and resilience in children with cancer and their parents that can be easily and widely disseminated.

DETAILED DESCRIPTION:
Childhood cancer patients and their parents are faced with significant stress at the time of diagnosis, during treatment, and over the course of recovery. The stress of cancer and its treatment can lead to significant emotional distress for many families. However, most families do not have access to programs that offer support for coping with cancer-related stress. The proposed work will address this gap by testing of the possible benefits of a novel internet delivered program to support children with cancer and their parents in coping with and communicating about a child's cancer. This online program includes modules to teach parenting, communication and coping skills to parents of children with cancer, and coping skills to their children who have been recently diagnosed with cancer. The research team includes experts from Vanderbilt University and Nationwide Children's Hospital with experience in pediatric oncology; stress, coping, and family communication in pediatric cancer; internet interventions in pediatric populations; and family-focused interventions to build coping and parenting skills. The study will test the effects of this program in 150 families of children with newly diagnosed cancer on reducing emotional distress up to 12 months after participation in the program. This project has the potential to lead to an evidence-based program to improve quality of life and resilience in children with cancer and their parents that can be easily and widely disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Child from ages 10 to 17 years old who has been diagnosed with cancer

Exclusion Criteria:

* Significant intellectual disability that would interfere with completing the online program

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Total Behavior Problems on the Child Behavior Checklist from baseline to 6 months | The Child Behavior Checklist will be completed near the time of entry into the study and repeated at 6 month follow ups
  Change in parents' report on the Child Behavior Checklist (a measure of their children's total emotional and behavioral problems).
Change in Total Behavior Problems on the Youth Self Report from baseline to 6 months | This measure will be completed near the time of entry into the study and repeated at 6 month follow ups
  Change in children's report on the Youth Self Report (a measure of their children's total emotional and behavioral problems).

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States